CLINICAL TRIAL: NCT03893474
Title: Quality-Assured Follow-up of Quiescent Neovascular Age -Related maculaR dEgeneration by Non-medical Practitioners: a Randomised Controlled Trial
Brief Title: Quality-Assured Follow-up of Quiescent Neovascular Age -Related maculaR dEgeneration by Non-medical Practitioners
Acronym: FENETRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Newcastle University (Other); Cardiff University (Other); City, University of London (Other); King's College London (Other); Manchester University NHS Foundation Trust (Other Government); University Hospitals Bristol and Weston NHS Foundation Trust (Other); York Teaching Hospitals NHS Foundation Trust (Other); Leeds Teaching Hospital NHS Foundation Trust (Unknown); Bradford Teaching Hospitals NHS Foundation Trust (Other Government); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BALK1005
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: AMD
Keywords: AMD; nAMD
MeSH Terms: interventions — Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Other): All investigations are the same in both arms, but patients within this arm will be seen in the hospital as per standard practice.
  Interventions: Diagnostic Test: OCT; Diagnostic Test: Visual Acuity
- Study Arm (Other): All investigations are the same in both arms, but patients within this arm will be seen in a community optometrist practice.
  Interventions: Diagnostic Test: OCT; Diagnostic Test: Visual Acuity

INTERVENTIONS:
Diagnostic Test: OCT — Optical Coherence Tomography of study eye.
Diagnostic Test: Visual Acuity — Visual acuity measured by ETDRS

SUMMARY:
This is a prospective, randomised, multi-site clinical trial testing the non-inferiority of community optometry follow-up of participants with QnAMD over 12 months

DETAILED DESCRIPTION:
Neovascular Age-Related Macular Degeneration (nAMD) is a common vision threatening condition affecting mainly patients over the age of 65. At some point during follow-up the disease becomes inactive in many cases and does not need more injections. The risk of a flare-up is high, however, and patients need to continue to be seen every month for a significant period of time.

Hospital-based eye clinics are struggling to cope with current and expected workload for assessing and treating patients with nAMD. Transferring care of these patients to the community closer to home would ease the workload for hospital based clinics and offer a better experience of care to patients.

This study will recruit 742 patients with nAMD who have reached this inactive phase of the disease. Half of the patients that want to take part will continue to have their follow-up appointments in the hospital eye clinics as usual. The other half, chosen by chance, will have follow-up visits every month in a community optometrist practice by trained optometrists. The research team will provide the training for community optometrists.

The study will seek to show that the community based care is no less safe than hospital-based care.

The study will also check what is the impact of this different way of offering care on the NHS budget and how the patients and practitioners perceive this. The study will involve several hospital eye clinics across the country and several community optometrist practices. Meetings will also be held with patients to discuss their priorities and needs when looking at how to set up the community based eye clinics.

During meetings with patients in preparation for this research, they felt positively about the possibility to receive care closer to home.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving treatment in nAMD injection clinics, who have reached the agreed definition of disease quiescence
* Informed consent
* Aged > 55 years
* Ability to perform study specific procedures

Exclusion Criteria:

* Significant media opacities (cataract, vitreous opacities) that would not allow good quality fundus imaging.
* Diabetic retinopathy of severity worse than mild non-proliferative stage and with any degree of diabetic maculopathy
* History of other causes of Choroidal Neovascularisation (myopic, angioid streaks, inflammatory, retinal dystrophies, secondary to Central Serous Chorioretinopathy, idiopathic).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 742 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of Participants who reactivate within 12 months of randomisation but are not identified as having re-activated (false negatives). | 12 months
  The proportion of Participants who reactivate within 12 months of randomisation but are not identified as having re-activated (false negatives).
Primary economic outcome: Incremental cost per quality adjusted life year (QALY) gained over the estimated patient lifetime estimated from an economic model informed by trial data. | 12 months
  Primary economic outcome: Incremental cost per quality adjusted life year (QALY) gained over the estimated patient lifetime estimated from an economic model informed by trial data.

SECONDARY OUTCOMES:
Diagnostic accuracy of the intervention (community optometry follow up of QnAMD) against the reference standard (rate of false negatives and false positives) | 12 months
  Diagnostic accuracy of the intervention (community optometry follow up of QnAMD) against the reference standard (rate of false negatives and false positives)
Rate of over-referral (i.e. Reference Standard is quiescent but classification is 'reactivated' or 'suspicious') | 12 months
  Rate of over-referral (i.e. Reference Standard is quiescent but classification is 'reactivated' or 'suspicious')
Mean change in visual acuity (measured with habitual correction and pinhole) for in the Participants intervention and control groups | 12 months
  Mean change in visual acuity (measured with habitual correction and pinhole) for in the Participants intervention and control groups
Rate of 'suspicious' lesion classification in community care | 12 months
  Rate of 'suspicious' lesion classification in community care
Rate of patient non-attendance and loss to follow up in secondary and primary care | 12 months
  Rate of patient non-attendance and loss to follow up in secondary and primary care
Use of health services and patient costs collected via eCRF and participant completed questionnaires | 12 months
  Use of health services and patient costs collected via eCRF and participant completed questionnaires
Costs of interventions and subsequent care to the NHS modelled over the estimated lifetime | 12 months
  Costs of interventions and subsequent care to the NHS modelled over the estimated lifetime
Modelled estimates of visual impairment and QALYs based on responses to the EQ-5D-5L. | 12 months
  Modelled estimates of visual impairment and QALYs based on responses to the EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Balaskas, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Derived] Vougioukalou S, Read SM, Csontos JK, Jones A, Jaber A, Sharma A, Balaskas K. Comparing community-based monitoring to hospital-based care of patients with quiescent age-related macular degeneration: a qualitative study of patient and practitioner perspectives on acceptability and access. BMJ Open. 2026 Feb 4;16(2):e101379. doi: 10.1136/bmjopen-2025-101379. PMID 41638748
- [Derived] Learoyd AE, Tufail A, Bunce C, Keane PA, Kernohan A, Robinson E, Jaber A, Sadiq S, Harper R, Lawrenson J, Vale L, Waterman H, Douiri A, Balaskas K; FENETRE study group. FENETRE study: quality-assured follow-up of quiescent neovascular age-related macular degeneration by non-medical practitioners: study protocol and statistical analysis plan for a randomised controlled trial. BMJ Open. 2021 May 11;11(5):e049411. doi: 10.1136/bmjopen-2021-049411. PMID 33980536